CLINICAL TRIAL: NCT05207410
Title: Effectiveness of Teaching Program for the Management of Upper GI Bleeding in Terms of Gain in Nurses' Knowledge and Practice
Brief Title: Effectiveness of Teaching Program for the Management of Upper GI Bleeding
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Shashi Prakash, Pursuing Postgraduate in Gastroenterology Nursing, Institute of Liver and Biliary Sciences, India
Other Study IDs: ILBS-UGIBCLD-100
Record Dates: First submitted 2021-12-27; First posted 2022-01-26 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Nurse
Keywords: Effectiveness; management of upper GI bleeding; planned teaching program; response time; nurses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 16 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A study to assess the effectiveness of teaching program for the management of upper GI bleeding in terms of gain in nurses' practice and knowledge related to management of upper GI bleeding among chronic liver disease patients visiting Emergency Room at ILBS, New Delhi.

The study assumes that- The nurses are practising as per their usual nursing practices while managing the patients with upper GI bleeding.

Nursing Personnel have some knowledge in the practice related to management of upper GI bleeding among CLD patients.

The nurses are documenting their nursing intervention correctly. The patient is managed by the nurses through a nursing team approach. (Any nursing professional from the nursing team can attend to the patient in the emergency room.) Structured teaching program will enhance the patient care related to the management of upper GI bleeding among chronic liver disease patients visiting Emergency Room.

The study hypothesis is tested at 0.05 level of significance: - H1 - There is a significant difference between mean knowledge score of nurses' before and after administration of Structured teaching Program as measured by Structured Questionnaire H2 - There is a significant difference between mean practice score of nurses' before and after administration of Structured teaching Program as measured by observation checklist H3 - There is a significant difference between mean practice response time score of nurses' before and after administration of Structured teaching Program as measured by observation checklist H4 - There is a significant association between nurses' knowledge and selected demographic and clinical variables of the patients visiting Emergency Room.

DETAILED DESCRIPTION:
A study to assess the effectiveness of teaching program for the management of upper GI bleeding in terms of gain in nurses' knowledge and practice related to management of GI bleeding among chronic liver disease patients visiting Emergency Room at ILBS, New Delhi.

The objectives of the study To determine the nurses' knowledge in the management of upper GI bleeding among chronic liver disease patients visiting Emergency Room before and after the administration of the structured teaching programme.

To determine the nurses' practices and nurses practice response time in the management of upper GI bleeding among chronic liver disease patients visiting Emergency Room before and after the administration of the structured teaching programme.

To assess the factors affecting the nurses' practice in the management of upper GI bleeding among chronic liver disease patients visiting emergency room.

To find out the association between nurses' knowledge in the management of upper GI bleeding among chronic liver disease patients visiting emergency room and the selected demographic variables of the nurses' working in emergency room.

Operational definition Assess: In this study it refers to evaluating the effectiveness of nurses' practice and related factors in the management of upper GI bleeding among chronic liver disease patients visiting Emergency Room.

Effectiveness: In this study, it refers to the power of nursing structured teaching program to bring about the changes in the nurses' practices measured by significant gain in knowledge score and assessed by structured knowledge questionnaire.

Nurse: In this study, it refers to the staff nurses as well as team leader on duty who are actively involved in direct care of CLD patients visiting emergency room with upper GI bleeding.

Practice: In this study, it refers to the performance of requisite interventions by the nurses related to management of upper GI bleeding among chronic liver disease patients visiting Emergency Room as measured by observation checklist.

Knowledge: In this study, it refers to the ability of nurses to respond correctly to structured knowledge questionnaire containing knowledge items on management of upper GI bleeding among CLD patients, as evident from knowledge scores.

Response time: In this study, it refers to the time from the arrival of the patient at Emergency Room gate till the patient gets a response from the emergency room nursing staff in term of implementing requisite nursing intervention(s) in the management of upper GI bleeding.

Factors- In this study, it refers to all those elements in the emergency room and characteristics of nurses that may influence the nurse's practice in providing quality care to CLD patients visiting Emergency Room with upper GI bleeding and includes their age, experience, nurse patient ratio, shift duration, emergency training, physical training, administrative policies, education level, knowledge, length of work.

Upper GI bleeding - In this study, it refers to classic upper GI bleeding symptoms or the history of recent upper GI bleeding for which a chronic liver disease patient visits the emergency room of ILBS.

Management of upper GI bleeding - In this study, it refers to all nursing intervention towards assessment of early initiation of clinical care and symptom management within the emergency room and includes the following: -

* Primary assessment,
* Resuscitation/stabilisation,
* History collection& health assessment,
* Supportive treatment,
* Transfer and referral. Chronic liver disease - In this study, it refers to patients diagnosed with Chronic liver disease and admitted in the emergency room for the management of upper GI bleeding.

Patients - In this study, it refers to the person either male or female who is coming for the management of upper GI bleeding among chronic liver disease patients visiting Emergency Room of ILBS hospital during the time of data collection Emergency Room (ER) -In this study, it refers to the emergency room of ILBS, New Delhi.

Structured Teaching Program - In this study, it refers to the structured teaching program designed by the researcher for the management of upper GI bleeding among chronic liver disease patients visiting Emergency Room and comprises of a checklist and guidelines.

Event - In this study, it refers to the visits made by a CLD patients with upper GI bleeding to the Emergency department of ILBS from 8 AM to 8 PM Assumptions The study assumes that- The nurses are practising as per their usual nursing practices while managing the patients with upper GI bleeding.

Nursing Personnel have some knowledge in the practice related to management of upper GI bleeding among CLD patients.

The nurses are documenting their nursing intervention correctly. The patient is managed by the nurses through a nursing team approach. (Any nursing professional from the nursing team can attend to the patient in the emergency room.) Structured teaching program will enhance the patient care related to the management of upper GI bleeding among chronic liver disease patients visiting Emergency Room.

Ethics Committee Clearance The Institutional Review Board clearance was obtained by two processes, Scientific Review Committee and Ethics Committee Clearance was obtained from Scientific Review Committee and Ethics Committee of College of Nursing, ILBS, and New Delhi.

Ethics approval to conduct the study was obtained from the college of nursing. All procedures to be performed in this study involving human participants are in accordance with the ethical standards of the Institutional Ethical Committee as laid down by WHO, ICMR and its later amendments. Informed Consent will be taken from each participant after explanation and giving Information Sheet Materials and Methods: - Quantitative research approach is used. Research Design in the study One group Pre test - Post test design is used

The symbols used means:

O1: Assessment of nurses' practices related to management of upper GI bleeding among CLD patients before intervention.

O2: Assessment of nurses' knowledge related to management of upper GI bleeding among CLD patients before intervention.

O3: Assessment of nurses' practices related to management of upper GI bleeding among CLD patients after intervention.

O4: Assessment of nurses' knowledge related to management of upper GI bleeding among CLD patients after intervention.

X: Structured teaching program The present study will be conducted in Emergency Room at ILBS hospital. In the present study, population comprises of Nurses working at ILBS. and the target population comprises of Nurses working in Emergency Room, and accessible population comprises of Nurses' providing care to upper GI bleeding among CLD patients visiting Emergency Room at the time of data collection.

Sample Size:

Nurses: Total Enumeration. [ 20 nurses} Events: Total Enumeration (Total number of events in the morning, evening and night shifts during data collection period will be observed i.e., 35 events).

Source of data Data will be collected from the study participants, nurses' record and observation method The variables used in this study is Research variables i.e. Independent Variable: Structured teaching program

Dependent Variable:

Knowledge of nurses regarding management of upper GI bleeding. Practices of nurses and their response time regarding management of upper GI bleeding.

Factors affecting nurses' practices in the management of upper GI bleeding among chronic liver disease patients.

Sociodemographic variables of nurses. Process of Data Collection For the final study, the data was collected in the month of November, 2021 in the Emergency Room, ILBS, New Delhi. Formal permission will be obtained from concerned authority to conduct the study. CLD patients who are coming to emergency unit with upper GI bleeding. Observation of nurses' practice were done by observation checklist from the time of receiving the patients from the entrance of emergency unit till the referral to endoscopy or ward/ICU for further management. Total enumeration sampling technique was used and those nursing personnel who will meet the selection criteria will be recruited. Participant information sheet will be provided to each participant to read followed by clear explanation of their rights and clarification of their queries. Informed consent was signed and taken from every participant.

During data collection period, nursing personnel was asked to fill their demographic profile data. Then principal investigator had assessed their practice using observation checklist followed by assessment of knowledge using structured knowledge questionnaire. The structured teaching programme was administered to nursing personnel in a group of 3 to 4 person. After administration of teaching programme, principal investigator reassessed the practice and knowledge of nursing personnel.

Tool for Data Collection:

These tools was selected after extensive review of literatures and expert's guidance.

Tool 1: Structured questionnaire to assess the Part-1: selected Socio-Demographic profile Part-2: knowledge of Nurses' regarding management of upper GI bleeding Part-3: factors affecting nurses' practices in the management of upper GI bleeding among chronic liver disease patients visiting Emergency Room.

Tool 2: Observation checklist with response time to assess the nurses' practice while managing patient with upper GI bleeding among chronic liver disease patients visiting emergency room.

ELIGIBILITY:
Inclusion Criteria:

* Nurses' who are involved in direct patient care and include the staff nurses' as well as team leader on duty.

Exclusion Criteria:

* Nurses' who are on long leave.
* Nurses who are on relieving duty. (pull out shift)

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The staff nurses as well as team leader on duty who are actively involved in direct care of CLD patients visiting emergency room with upper GI bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Knowledge of Nurses' in the management of upper GI bleeding among chronic liver disease patients visiting Emergency Room. | up to 5 weeks
  Structured knowledge questionnaire to assess nurses' knowledge regarding upper GI bleeding. It consists of 30 multiple choice knowledge questionnaire with minimum 0 and maximum 30 marks and higher score means better result.
Practice of Nurses' in the management of upper GI bleeding among chronic liver disease patients visiting Emergency Room. | up to 5 weeks
  Observation Checklist for the assessment of Practice of Nurses regarding upper GI bleeding The performance of activity is awarded a score of 'One' and non-performance is awarded a score of 'Zero'. The maximum possible score is 34 and minimum 0 and higher score means better result.

CONTACTS AND LOCATIONS:
Overall Officials: Shashi Mr Prakash, Nursing, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India